CLINICAL TRIAL: NCT01382745
Title: A Phase II Clinical Study Using Nimotuzumab in Combination With External Beam Radiation Therapy in the Treatment of Patients With Carcinomas of the Anal Canal
Brief Title: Nimotuzumab With Radiotherapy in the Treatment of Anal Canal Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Dr. Te Vuong (Other)
Collaborators: YM BioSciences (Industry)
Responsible Party: Sponsor-Investigator, Dr. Te Vuong, MD-Director Radiation Oncology, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-044
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Squamous Cell Carcinoma of Anal Canal
MeSH Terms: interventions — nimotuzumab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab (Experimental): Patients will receive weekly injections of Nimotuzumab (200mg/injection) for 12 weeks and standard external beam radiotherapy
  Interventions: Drug: Nimotuzumab; Radiation: Intensity Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Drug: Nimotuzumab — 200mg Nimotuzumab once a week for 12 weeks
Radiation: Intensity Modulated Radiation Therapy (IMRT) — IMRT radiation therapy with doses varying from 45Gy-54Gy in 25-30 fractions

SUMMARY:
The objective of this study is to demonstrate the feasibility of using Nimotuzumab and radiation in the treatment of squamous cell carcinomas of the anal canal in order to achieve a 65% local control rate with a better toxicity profile than the conventional treatment. Patients with high toxicity risks (HIV+ and fragile patients) will be selected for this study.

ELIGIBILITY:
Inclusion Criteria:

For both step I and II:

* Patients with histologically confirmed squamous cell carcinoma of the anal canal
* Aged 18 years or older
* ECOG: 0-1-2
* Adequate contraception in women of child-bearing potential and for men
* Ability to understand and the willingness to sign a written informed consent document.
* HIV-positive patients with T1-2 anal canal tumors, or
* Patients with anal canal tumors not eligible for conventional chemotherapy (for example, due to age and/or co-morbidities)
* Patients who have already started radiotherapy for anal canal cancer

For step II:

* HIV-positive patients with T1, T2 anal canal tumors
* HIV-negative patients not eligible for conventional chemotherapy (for example, due to age and/or co-morbidities)
* HIV-negative patients with T1-2 anal canal cancer

Exclusion Criteria:

For both step I and II:

* Patients receiving any other investigational agents
* Previous treatment with anti-EGFR drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Nimotuzumab or other agents used in study.
* Previously treated with pelvic radiotherapy.
* Lesions not suitable for radiotherapy
* Patients with uncontrolled hypercalcemia
* Uncontrolled intercurrent illness
* Pregnant or breast-feeding women
* Any concurrent active malignancy
* Patients with T3-4 anal canal tumors or patients with nodes positive.

Step I:

* HIV-negative patients with anal canal tumors that are judged suitable for current treatment consisting in radiotherapy and 5-FU and MMC chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-01; Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 1 month post end of treatment
  Toxicity evaluation will include all toxicities occurring while the patient is receiving treatment, and will be monitored using the CTCAE guide version 3.0.
Local tumor response rate | 8 weeks post end of radiation treatment
  Tumor response rates will be evaluated using the MRI performed at 8-weeks post end of radiotherapy treatment.

SECONDARY OUTCOMES:
Overall cancer-free survival | 5 years post end of treatment
Overall survival | 5 years post end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Te Vuong, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada